CLINICAL TRIAL: NCT04131621
Title: A Phase II, Open-label, Non-randomized, Multi-center Study Evaluating the Efficacy and Safety of Nivolumab Plus Ipilimumab in Patients With Cancer of Unknown Primary Site Who Are Relapsed After or Refractory to Platinum-based Chemotherapy
Brief Title: Nivolumab/Ipilimumab in Second Line CUP-syndrome
Acronym: CheCUP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Alwin Kraemer, Prof. Dr. med., University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-8WY
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Cancer of Unknown Primary Site
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab/Ipilimumab (Experimental)
  Interventions: Biological: Nivolumab/Ipilimumab

INTERVENTIONS:
Biological: Nivolumab/Ipilimumab — Immune checkpoint inhibitor combination

SUMMARY:
To compare the efficacy of nivolumab plus ipilimumab in subjects with high vs. Intermediate/low TMB poor-prognosis CUP (non-specific subset) who are relapsed or refractory to platinum-based first-line chemotherapy.

To evaluate the efficacy of nivolumab plus ipilimumab in subjects with poor-prognosis CUP (non-specific subset) who are relapsed or refractory to platinum-based first-line chemotherapy

ELIGIBILITY:
Inclusion Criteria

* Signed Informed Consent Form
* Able and willing to comply with the study protocol
* Age ≥ 18 years at time of signing Informed Consent Form
* Histologically-confirmed disseminated or advanced unresectable CUP diagnosed according the criteria defined in the 2015 ESMO Clinical Practice Guidelines for CUP. Acceptable disease histology includes:

  * Adenocarcinoma of unknown primary site (ACUP)
  * Poorly differentiated adenocarcinoma of unknown primary site
  * Poorly differentiated carcinoma of unknown primary site
  * Squamous cell carcinoma of unknown primary site (SCUP)
* At least one lesion that is measurable according to RECIST v1.1
* Availability of a tumor FFPE block either fresh or archival if obtained ≤ 6 months at Screening that is sufficient for generation of a TruSight Oncology 500 (TSO500) panel at the central reference pathology laboratory
* Availability of test reports confirming local CUP diagnosis. If test reports confirming local CUP diagnosis are not available, an FFPE block must be submitted that is sufficient to allow for central confirmation of CUP diagnosis
* Disease relapse or progression after at least three cycles of a platinum-based standard chemotherapy. There is no upper limit of prior treatments received.
* ECOG performance status of 0 - 2
* Life expectancy ≥ 12 weeks
* Eligible for immune checkpoint inhibitor
* Adequate hematologic and end-organ function
* For women of childbearing potential and men capable of reproduction: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 5 months for women and 7 months for men, respectively after the last dose of study treatment.
* Recovery from significant toxicity from platinum-doublet therapy to Grade ≤ 1, except for alopecia and for neurosensory toxicity, which must be ≤ 2
* Recovery from active infections requiring intravenous antibiotics, with antibiotic therapy ceased for ≥ 7 days prior to planned start of therapy

Exclusion Criteria

* Subjects with any of the specific non-CUP neoplasms identified in the ESMO CUP guidelines, including:

  * Non-epithelial cancer
  * Extragonadal germ-cell tumor
* Subjects belonging to any of the following subsets of CUP with favorable prognoses:

  * Poorly differentiated carcinoma with midline distribution
  * Women with papillary adenocarcinoma of the peritoneal cavity
  * Women with adenocarcinoma involving only the axillary lymph nodes
  * Squamous cell carcinoma restricted to cervical lymph nodes
  * Poorly and well differentiated neuroendocrine tumors
  * Men with blastic bone metastases and elevated PSA
  * Subjects with a single, small tumor potentially resectable and/or amenable to radiotherapy with curative intent
  * Colon cancer-type CUP
* Known presence of brain or spinal cord metastasis (including metastases that have been irradiated), as determined by CT or magnetic resonance imaging (MRI) evaluation during screening
* History or known presence of leptomeningeal disease
* Uncontrolled or symptomatic hypercalcemia (serum calcium ≥ 2.9mmol/L)
* Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including active viral or other hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus (HIV) infection
* Positive for hepatitis C virus (HCV) infection at screening
* Positive for hepatitis B surface antigen (HBsAg) at screening
* Active tuberculosis at Screening
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia (including active ventricular arrhythmia requiring medication), or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy other than CUP within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Known allergy or hypersensitivity to any component of the immunotherapy, including history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins and to Chinese hamster ovary cell products or other recombinant human or humanized antibodies for nivolumab and ipilimumab.
* Subjects with an active, known or suspected autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, myocarditis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents, or other immuno-suppressive medications within 14 days of study treatment. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents for adults, or > 0.25 mg/kg daily prednisone equivalent for adolescents are permitted, in the absence of active autoimmune disease.
* Subjects who received prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 5) or baseline before administration of study drug. Subjects with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum based therapy, are permitted to enroll.
* Treatment with any chemotherapy, radiation therapy, biologics for cancer, or investigational therapy within 28 days of first administration of study treatment (subjects with prior cytotoxic or investigational products < 4 weeks prior to treatment initiation might be eligible after discussion between investigator and sponsor, if toxicities from the prior treatment have been resolved to Grade 1 (NCI CTCAE version 5).
* Subjects must not have received a live / attenuated vaccine within 30 days of first treatment.
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the last dose of study treatment or intention of fathering a child within 7 months after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 months
  Months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Pouyiourou M, Kraft BN, Wohlfromm T, Stahl M, Kubuschok B, Loffler H, Hacker UT, Hubner G, Weiss L, Bitzer M, Ernst T, Schutt P, Hielscher T, Delorme S, Kirchner M, Kazdal D, Ball M, Kluck K, Stenzinger A, Bochtler T, Kramer A. Nivolumab and ipilimumab in recurrent or refractory cancer of unknown primary: a phase II trial. Nat Commun. 2023 Oct 24;14(1):6761. doi: 10.1038/s41467-023-42400-5. PMID 37875494